CLINICAL TRIAL: NCT06887413
Title: TACTIC Coronary Thrombus Aspiration With Cath Rx In Anterior Myocardial Infarction: A Randomized Control Trial.
Acronym: TACTIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC
Record Dates: First submitted 2025-03-04; First posted 2025-03-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anterior Myocardial Infarction
Keywords: STEMI; thromboaspiration; anterior myocardial infarction; INDIGO CAT RX; indigo system; HEART ATTACK
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects randomized to the control arm will be treated with standard PPCI (No Intervention): Subjects randomized to the control arm will be treated with standard PPCI
- - Treatment arm: Subjects randomized to the treatment arm will be treated with the CAT RX (Experimental): Treatment arm: Subjects randomized to the treatment arm will be treated with the CAT RX
  Interventions: Procedure: THROMBOASPIRATION WITH INDIGO SYSTEM

INTERVENTIONS:
Procedure: THROMBOASPIRATION WITH INDIGO SYSTEM — Subjects randomized to the treatment arm will be treated with the CAT RX as previously described.
  Arms: - Treatment arm: Subjects randomized to the treatment arm will be treated with the CAT RX

SUMMARY:
The aim of this study is to evaluate the impact of sustained thrombectomy with INDIGO ASPIRATION SYSTEM using CAT RX versus no thrombectomy during primary percutaneous coronary intervention (PPCI) on microvascular obstruction and infarct size, as measured by cardiovascular magnetic resonance (CMR) between 3 and 5 days post PPCI, in patients with anterior STEMI

DETAILED DESCRIPTION:
Prospective, randomized 1:1, controlled, open label, multicentred, investigator initiated clinical investigation in 14 European sites. 140 patients will be enrolled in the study after coronary angiography confirming prox or mid LAD occlusion. Patients will be randomised in one of the following arms:

Treatment arm: Subjects randomized to the treatment arm will be treated with the CAT RX as previously described.

Control arm: Subjects randomized to the control arm will be treated with standard PPCI .

Participants will undergo a cardiac MRI, including gadolinium contrast imaging, within 3-5 days following the index procedure. If clinical contraindications prevent the MRI from being performed within this timeframe, it should be conducted as soon as the participant is clinically stable.

After the discharge, In-person or phone follow-ups will take place at 30 days, and 12 months post-PCI.

Primary endpoint will be measured at 3-5 days post procedure where a microvascular obstruction will be assed by CMR mass.

Secondary endpoints will be assessed: Secondary CMR endpoint - measured at 3-5 days post PPCI:Infarct size, as a percent of LV mass

* Left ventricular end-systolic volume (LVESV)
* Left ventricular end-diastolic volume (LVEDV)
* Left ventricular end-systolic volume index
* Left ventricular end-diastolic volume index
* Ejection fraction (EF)

Secondary exploratory clinical and angiographic endpoint:

Measured at the end of the procedure:

* TIMI 3 flow at the end of primary PCI
* Post PCI non-hyperemic angio-derived IMR measurements. PCI

Measured at 1 year post procedure:

- MACE at 1-year follow-up (a composite end point of all-cause death, myocardial infarction, pMCS implant, target lesion revascularization, stent thrombosis, ICD implantation or HF hospitalizations) and each individual component.

Safety endpoint:

Measured at 1 month post procedure:

- Device-related SAE(s) and Stroke

ELIGIBILITY:
INCLUSION CRITERIA

1. Age >18 and <75 years old
2. Acute anterior STEMI with ≥2 mm in two (2) or more contiguous anterior leads or ≥4 mm total ST-segment deviation sum in the anterior leads V1-V4 AND anterior wall motion abnormality noted on a diagnostic quality left ventriculogram or echocardiogram
3. Culprit lesion proximal or mid LAD at coronary angiography
4. TIMI thrombus grading > 3 or TIMI flow 0 after guidewire crossing the lesion.
5. Patient presents to the hospital between 1 - 6 hours of ischemic pain onset
6. Patient indicated for primary percutaneous coronary intervention (PPCI)

EXCLUSION CRITERIA

1. Unable to give Informed consent.
2. Life expectancy < 1 year.
3. Contraindication to PCI
4. STEMI due to stent thrombosis
5. Spontaneous coronary aretery dissection
6. Patient undergone any kind of maneuvers to restore flow before randomization
7. Unwitnessed cardiac arrest OR ≥30 minutes of cardiopulmonary resuscitation (CPR) prior to enrolment OR any cardiac arrest with impairment in mental status, cognition or any global or focal neurological deficit
8. New onset of stroke symptoms and NIHSS >2, prior to index procedure
9. Known intolerance to aspirin, clopidogrel, ticagrelor, heparin, contrast media.
10. Active severe bleeding
11. Severe hepatic/kidney impairment
12. Administration of fibrinolytic therapy within 24 hours prior to enrolment
13. Cardiogenic shock defined as systemic hypotension (systolic BP <90 mmHg or the need for inotropes/pressors to maintain a systolic BP >90 mmHg), plus one (1) of the following: any requirement for pressors / inotropes prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion, or use of IABP or any other mechanical circulatory support device
14. Inferior STEMI or suspected right ventricular failure
15. Severe valvulopathy
16. Acute cardiac mechanical complication: LV-free wall rupture OR interventricular septum rupture OR acute mitral regurgitation

Medical Conditions & History:

1. Suspected or known pregnancy
2. Suspected systemic active infection
3. History or known hepatic insufficiency prior to catheterization
4. Undergoing a renal replacement therapy
5. Chronic obstructive pulmonary disease (COPD) with home oxygen therapy or on chronic steroid therapy
6. Contraindication to perform MRI or use gadolinium [creatinine clearance (CrCl) <30 mL/min, non-compatible implant, claustrophobia]

Cardiovascular history

1. Known or evidence of prior MI, including pathologic Q-waves in non-anterior leads
2. Prior coronary artery bypass graft surgery (CABG) or LAD PCI
3. History of heart failure (documented history of EF <40% or documented hospitalization for HF within 1 year prior to screening
4. Prior aortic valve surgery or TAVR
5. Left bundle branch block (new or old)
6. History of stroke/TIA within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Microvascular obstruction | Within 3-5 days post procedure
  Incidence of Microvascular obstruction (MVO) assessed by Cardiac Magnetic Resonance

SECONDARY OUTCOMES:
Secondary CMR endpoint: | Within 3-5 days post procedure
  Left Ventricular Mass in % Left ventricular end-systolic volume (LVESV) Left ventricular end-diastolic volume (LVEDV) Left ventricular end-systolic volume index Left ventricular end-diastolic volume index Ejection fraction (EF)
Secondary exploratory clinical and angiographic endpoint: | At the end of the procedure
  Incidence of TIMI 3 flow at the end of primary PCI Post PCI non-hyperemic angio-derived IMR measurements. PCI
Safety endpoint | At 1 year Follow Up
  Incidence of MACE at 1-year follow-up (a composite end point of all-cause death, myocardial infarction, pMCS implant, target lesion revascularization, stent thrombosis, ICD implantation or HF hospitalizations) and each individual component
Safety endpoint | At 1 month post procedure
  Incidence of device-related SAE(s) and Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Alaide Chieffo, Principal Investigator — San Raffaele Hospital
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Milani, Italy

IPD SHARING:
Plan to Share IPD: No